CLINICAL TRIAL: NCT06932822
Title: Mental Imagery to Enhance Procedural Skills in Peripheral Venous Catheterization: A Randomized Simulation Study in Medical Students
Brief Title: Mental Imagery to Enhance Procedural Skills in Peripheral Venous Catheterization
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Principal Investigator, Nicolas BOULET, Medical Doctor, Principal Investigator, Centre Hospitalier Universitaire de Nīmes
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MI-24.11.07
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Peripheral Venous Catheterization; Simulation Training; Mental Imagery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Insertion of a peripheral venous catheter on a simulation mannequin after theoretical video instruction
- Mental Imagery (Experimental): Insertion of a peripheral venous catheter on a simulation mannequin after theoretical video instruction and mental visualization session
  Interventions: Other: Mental Imagery

INTERVENTIONS:
Other: Mental Imagery — Placement of a peripheral venous catheter on a simulation mannequin after a mental visualization session
  Arms: Mental Imagery

SUMMARY:
Peripheral venous catheter insertion has a slow learning curve, and is rarely performed by medical students. Most medical interns do not master this procedure independently at the start of their residency.

It's a painful procedure for the patients, and therefore unsuitable for "in vivo" training at the patient's bedside For this type of procedure, it would appear necessary to develop alternative teaching methods, as well as pedagogical tools that can modify the learning curve to make it faster.

Mental imagery is a technique that involves creating vivid, detailed mental images in the mind. It is often used in a variety of contexts, such as mental preparation, stress management, learning or goal achievement Initially used in mental preparation for sports, it made its appearance as a pedagogical tool in the medical field in the 2010s, with several studies demonstrating its value in learning procedural gestures (training in laparoscopic surgery, cystoscopy).

The aim of our study is to investigate the impact of a mental imagery session on peripheral venous catheter placement success in 5th-year medical students, on a simulation mannequin.

ELIGIBILITY:
Inclusion Criteria:

* 5th-year medical student at the Nîmes medical school taking part in the peripheral venous catheter insertion training workshop
* No other conditions required.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
First puncture success rate | 30 minutes
  Successful peripheral venous catheterization on first puncture, with no complications

SECONDARY OUTCOMES:
Revised Mental Imagery Questionnaire (MIQ)-3 variation | 30 minutes
  Change in Revised MIQ-3 score (mental visualization performance score) before and after the workshop. From 7 to 56.
Revised Mental Imagery Questionnaire (MIQ)-3 comparison | 30 minutes
  Comparison of the revised Mental Imagery Questionnaire-3 score (mental visualization performance score) between "mental visualization" and "control" groups. From 7 to 56
Puncture number | 30 minutes
  Comparison of puncture number between groups
Procedure complications | 30 minutes
  Comparison of number of complications
  * Arterial puncture
  * Failure
  * Non-functioning IV infusion

IPD SHARING:
Plan to Share IPD: No